CLINICAL TRIAL: NCT04047979
Title: Systems Biology of Zoster Vaccine Recombinant, Adjuvanted (SHINGRIX)
Brief Title: Systems Biology of Zoster Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Nadine Rouphael, Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00105838; 1U19AI090023 (NIH)
Record Dates: First submitted 2019-08-06; First posted 2019-08-07 (Actual); Results first posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Zoster; Zoster Varicella; Shingles; Chicken Pox
Keywords: Zoster; Immune responses; Vaccine; Vaccine Trials; Clinical Trials; Chicken Pox; Shingles
MeSH Terms: conditions — Herpes Zoster; Chickenpox

STUDY DESIGN:
Intervention Model Description: Single center, open label mechanistic study in which older adult subjects will receive Zoster vaccine recombinant, adjuvanted Vaccination will occur on Day 0 and Day 60. There will be no randomization, study participant or clinical study personnel blinding, or masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Younger Group (Experimental): Participants between the ages of 50 to 60 years will receive two doses of Zoster vaccine recombinant, adjuvanted (Shingrix®)
  Interventions: Biological: Shingrix®
- Older Group (Experimental): Participants who are ≥70 year old will receive two doses of Zoster vaccine recombinant, adjuvanted (Shingrix®)
  Interventions: Biological: Shingrix®

INTERVENTIONS:
Biological: Shingrix® — A zoster vaccine recombinant, adjuvanted, recently approved by the FDA for prevention of herpes zoster (shingles) in adults aged 50 years and older. It is given in two doses (0.5 mL each): at 0 and 2 to 6 months.

SUMMARY:
The purpose of the study is to better understand how the immune system responds to the new herpes zoster (shingles) vaccine (Shingrix®). The study will be looking at certain markers in the blood after vaccination with Shingrix®.

DETAILED DESCRIPTION:
Varicella zoster virus (VZV) can cause two distinct diseases: chicken pox (varicella) and herpes zoster (shingles). The primary infection with VZV causes chicken pox, a widespread rash occurring with fever, mostly in childhood. The virus can then remain dormant in a person's body and has the ability to reactivate later in life causing shingles. Shingles is a painful rash, occurring mostly in older individuals or those who have a weakened immune system. After resolution of the rash, individuals may experience persistent pain in the same area, called post-herpetic neuralgia.

The purpose of the study is to better understand how the immune system responds to the new herpes zoster (shingles) vaccine (Shingrix®). In particular, looking at certain markers in the blood after vaccination with Shingrix®.

The study will be an open label clinical trial in healthy older adults. There will be two groups of participants: those aged 50 to 60 years or those who are 70 years old and above, both groups will receive the vaccine. This will help compare the immune response to the herpes zoster vaccine in different age cohorts of older adults.

Subjects will be recruited by flyer advertisements. Interested individuals will be screened for the study and if they qualify they will be consented and enrolled in the study. Blood samples will be collected and banked. There are optional storage of data/specimens for future research including: being contacted for future studies, having contact information and limited medical information entered into a clinic database, and storage of Protected Health Information and samples for future research (yes, no, and de-identified).

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be able to understand and provide informed consent.
2. Adults aged 50-60 years, or community dwelling adults aged 70 years and above.

Exclusion Criteria:

1. Inability or unwillingness of a subject to give written informed consent or comply with study protocol.
2. Receipt of immune products:

   * Receipt of blood products within 6 months prior of the first dose of the study Zoster vaccine or expected receipt through 6 months after vaccination with the second dose of the study Zoster vaccine.
   * Receipt of any vaccine within 4 weeks prior to vaccination with any of the two doses of the study Zoster vaccine or expected receipt within 4 weeks after vaccination with any of the two doses of the study Zoster vaccine.
   * Receipt of any Zoster or varicella vaccines at any time prior to study entry.
3. Subject taking any non-topical antiviral therapy with activity against herpes viruses, including but not limited to acyclovir, famciclovir, valacyclovir, and ganciclovir 3 days prior to each vaccination or 14 days after.
4. Prior history of shingles.
5. Presence of certain co morbidities or immunosuppressive states such as:

   * Chronic medical problems including (but not limited to) insulin-dependent diabetes, severe (at the discretion of the investigator or study physician) heart, lung, liver, or kidney diseases; auto immune diseases; severe gastrointestinal diseases; and uncontrolled hypertension.
   * Impaired immune function or chronic infections including (but not limited to) HIV, hepatitis B or C, tuberculosis, organ transplant, cancer, current and or expected receipt of chemotherapy, radiation therapy, steroids [i.e., > 20 mg of prednisone given daily or on alternative days for 2 weeks or more in the past 90 days); (nasal (less than 1mg/day of fluticasone equivalent inhaled corticosteroid is allowable) and topical steroids are allowed)], antitumor necrosis factor agents, or any other immunosuppressive therapy, anatomic or functional asplenia, congenital immunodeficiency.
6. Conditions that could affect the safety of the subjects such as:

   * Severe reactions to prior vaccinations.
   * History of anaphylactic/anaphylactoid reaction to any component of the vaccines.
   * History of bleeding disorders.
7. Any acute illness, including any fever (> 100.4 F [> 38.0 C], regardless of the route) within 3 days prior to study entry.
8. Social, occupational, or any other condition that in the opinion of the investigator might interfere with compliance with the study and vaccine evaluation.
9. Alcohol or drug abuse and psychiatric conditions that in the opinion of the investigator would preclude compliance with the trial or interpretation of safety or endpoint data.
10. Use of investigational drugs within 12 months of participation.
11. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator or study physician, may pose additional risks from participation in the study, may interfere with the subject's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.
12. Women of childbearing potential.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Rouphael, MD, Principal Investigator — Emory University
Locations (1):
- The Hope Clinic, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: At the time of publication or 9 months after submission of the manuscript. It will be available indefinitely.
Access Criteria: Data will be uploaded into www.immport.org and made available to researchers with a registered account.
  Type of Analysis: Any Purpose
  Mode of Access: Data will be shared on www.immport.org
URL: http://www.immport.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Younger Group | Older Group
Started | 30 | 8
Completed | 18 | 8
Not Completed | 12 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Younger Group | Older Group | Total
Number analyzed (Participants) | 30 | 8 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (2.9) | 71.0 (1.2) | 57.9 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 3 | 14
  Male | 19 | 5 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 30 | 8 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 2 | 17
  White | 15 | 6 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 8 | 38

OUTCOME MEASURES:

1. Primary Outcome: Change in Innate Immune Signatures Post-vaccine Dose
Description: Will be assessed between D0, D1, and D7 and each dose of Zoster vaccine recombinant, adjuvanted, in both age cohorts: 50-60 years and >70 years of age. Results will be reported using Mean Normalized Enrichment Score (NES) of the Antiviral Interferon Signature Module (NES reflects the degree to which the activity level of a set of transcripts is overrepresented at the extremes (top or bottom) of the entire ranked list of transcripts within a sample and is normalized by accounting for the number of transcripts in the set. An NES of 0 indicates no change from baseline, a negative score reflects a reduction in the score (less activity), and a positive score reflects more activity of the module).
Time Frame: Day 1 from Day 0, Day 7 from Day 0, Day 61 from day 60, Day 67 from day 60
Population: Population of the outcome differ per time point based on the Number of participants that completed each follow up.
Measure: Mean (Standard Deviation); unit: Normalized Enrichment Score (NES)
Arm/Group | Younger Group | Older Group
Number analyzed (Participants) | 27 | 8
Normalized Enrichment Score (NES)
  Innate Immune signature at Day 1 from Day 0 | 1.6801 (0.8987) | 2.096 (0.2983)
  Innate Immune signature at Day 7 from Day 0: number analyzed (Participants) | 26 | 8
  Innate Immune signature at Day 7 from Day 0 | -0.5609 (1.3293) | -1.1284 (1.1369)
  Innate Immune signature at Day 61 from Day 60: number analyzed (Participants) | 21 | 8
  Innate Immune signature at Day 61 from Day 60 | 2.096 (0.3645) | 1.9814 (1.1519)
  Innate Immune signature at Day 67 from Day 60: number analyzed (Participants) | 19 | 8
  Innate Immune signature at Day 67 from Day 60 | -0.0081 (1.3921) | -1.071 (1.1055)

2. Secondary Outcome: Safety of Zoster Vaccine Recombinant, Adjuvanted
Description: Differences in related adverse events and serious adverse events between each dose of Zoster vaccine recombinant, adjuvanted, in both age cohorts. Number of participants with related AEs and SAEs (assessed within 7 days post-vaccination) will be reported.
Time Frame: Day 270 post-intervention
Population: Population analyzed in this outcome includes participants that completed the last follow up at 270 days post-intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Younger Group | Older Group
Number analyzed (Participants) | 18 | 8
Participants
  Number of participants with AEs at Day 270 for First vaccine dose | 4 | 0
  Number of participants with SAEs at Day 270 for First vaccine dose | 0 | 0
  Number of participants with AEs at Day 270 for Second vaccine dose: number analyzed (Participants) | 17 | 8
  Number of participants with AEs at Day 270 for Second vaccine dose | 1 | 0
  Number of participants with SAEs at Day 270 for Second vaccine dose: number analyzed (Participants) | 17 | 8
  Number of participants with SAEs at Day 270 for Second vaccine dose | 0 | 0

ADVERSE EVENTS:
Time Frame: Throughout study duration, an average of 270 days.
Arm/Group | Younger Group | Older Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/30 | 1/8
Other Adverse Events (participants affected / at risk) | 7/30 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Younger Group (N=30) | Older Group (N=8)
Cerebrovascular ischemia (Nervous system disorders) | 0 (0) | 1 (1)
West Nile Virus (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Younger Group (N=30) | Older Group (N=8)
Peripheral Neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Vertigo (General disorders) | 1 (1) | 0 (0)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ureteroscopy with lithotripsy (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertension emergency (Cardiac disorders) | 1 (1) | 0 (0)
Allergic rhinitis (General disorders) | 1 (1) | 0 (0)
Automobile accident (General disorders) | 1 (1) | 0 (0)
Reconstructive surgery 3rd, 4th, 5th phalange (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/79/NCT04047979/Prot_SAP_001.pdf
  • Informed Consent Form (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/79/NCT04047979/ICF_000.pdf